CLINICAL TRIAL: NCT04814693
Title: A Prospective, Post-Market, Multicenter, Randomized Controlled Trial to Compare the Performance of the EndoRotor® System Versus Conventional Endoscopic Techniques for Direct Endoscopic Necrosectomy of Walled Off Necrosis - The RESOlVE Trial
Brief Title: Conventional Endoscopic Techniques Versus EndoRotor® System for Necrosectomy of Walled of Necrosis
Acronym: RESOlVE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Interscope, Inc. (Industry)
Responsible Party: Principal Investigator, Marco J. Bruno, Prof. Marco Bruno, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-0061
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Acute Pancreatitis; Necrosis; Pancreas, Acute (Infectious)
MeSH Terms: conditions — Pancreatitis; Necrosis; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Subjects in this study will be included in either the intervention arm (EndoRotor) of control arm (conventional procedures).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional arm (Experimental): Subjects randomized to the control device arm will undergo treatment with the EndoRotor System, which is a powered debridement tool intended for use in endoscopic procedures to resect and remove necrotic debris during direct endoscopic necrosectomy (DEN) for walled-off necrosis. The system consists of capital components including a power console, roll stand, vacuum pump, and foot control; as well as disposable components including a single-use catheter, purge kit, and suction bag. The EndoRotor System has CE-Mark 613797 and is cleared for use by the FDA in the United States.
  Interventions: Device: EndoRotor® System (Interscope, Inc., Northbridge, MA USA),
- Control arm (Active Comparator): Subjects randomized to the control device arm will undergo conventional DEN as per the standard of care. Investigators will choose conventional DEN instruments according to their preference.
  Interventions: Procedure: Conventional endoscopic devices (according to standards of care)

INTERVENTIONS:
Device: EndoRotor® System (Interscope, Inc., Northbridge, MA USA), — The EndoRotor System is intended for use in endoscopic procedures to resect and remove necrotic debris during DEN for WON. DEN with the EndoRotor System (study device) is considered to be standard of care therapy for patients with WON and not investigational.
  Arms: Interventional arm
Procedure: Conventional endoscopic devices (according to standards of care) — Endoscopic devices used to perform conventional DEN will be chosen according to standard of care and Investigator preference.
  Arms: Control arm

SUMMARY:
In acute pancreatitis, approximately 20% of the cases result in severe necrotizing pancreatitis which is associated with significant morbidity and mortality. Necrotizing pancreatitis is characterized by the development of an acute necrotic collection and as this collection persists beyond 4 weeks, walled off necrosis (WON) encapsulates the collection. To date, this is treated by the step-up approach, which contains percutaneous drainage and minimally invasive video assisted retroperitoneal debridement (VARD) or endoscopic ultrasound (EUS) guided drainage followed by direct endoscopic necrosectomy (DEN). Different DEN techniques are available for the treatment of WON, however, there is a lack of effective endoscopic instruments to perform DEN. Recently, the first dedicated alternative to conventional DEN has been cleared for use, namely the EndoRotor® Resection System. This device is a powered mechanical debridement device intended for use in endoscopic procedures to resect and remove necrotic debris during DEN for WON. Previous (pilot and feasibility) studies showed promising results in terms of the amount of procedures, adverse events and length of hospital stay.

Therefore, aim of this study is to assess the performance of the EndoRotor, as compared to conventional endoscopic techniques, for direct endoscopic necrosectomy (DEN) of walled off necrosis (WON) in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic pancreatic necrosis due to acute pancreatitis that have an indication to undergo endoscopic necrosectomy after having undergone EUS-guided drainage.

  a. Stent must be in place for a minimum of 2 days prior to the DEN procedure.
* Patients who can tolerate repeat endoscopic procedures.
* Subjects with the ability to understand the requirements of the study, who have provided written informed consent, and who are willing and able to return for the required follow-up assessments.
* ASA classification < 5.

Exclusion Criteria:

* Documented pseudoaneurysm > 1 cm within the WON.
* Subject unable or unwilling to provide informed consent.
* Intervening gastric varices or unavoidable blood vessels within the WON access tract (visible using endoscopy or endoscopic ultrasound).
* Coagulation disorders or anti-coagulant therapy which cannot be discontinued (aspirin allowed).
* Any condition that in the opinion of the Investigator would create an unsafe clinical situation or stent placement that would not allow the patient to safely undergo an endoscopic procedure.
* Pregnant or lactating women or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator, and/or are not willing to use reliable contraception for the duration of study participation.
* Patient is enrolled in another trial that could interfere with the endpoint analyses of this trial.
* Prior necrosectomy on existing collection.
* Greater than 2 pancreatic / extra-pancreatic fluid collections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
The number of DEN procedures required to achieve resolution of WON | During a 6 month follow up period
  1. Resolution is defined as clinical improvement of WON symptoms precluding the need for additional endoscopic or surgical interventions.
  2. Clinical improvement is defined according to the criteria used in the PANTER trial and TENSION trial.8,15 "Clinical improvement" was defined as:
  i. Improved function of at least two organ systems (i.e. circulatory, pulmonary, renal) according to the Investigator's medical judgement within 72 hours, or; ii. At least 10% improvement of two out of three parameters of infection (i.e. C-reactive protein, leucocyte count or temperature) within 72 hours.

SECONDARY OUTCOMES:
Adverse events | During a 6 month follow up period
  The occurrence of all adverse events measured from the Index Procedure through the 6 Month Post Necrosectomy Follow-up Visit
Conversion to surgery defined as number of subject that require surgical intervention as a result of DEN failure as assessed by the Investigator during the index procedure through the 6 month post necrosectomy follow-up visit | During a 6 month follow up period
  In case of conversion to surgery, reason for conversion and type of surgical procedure
Length of hospitalization | During a 6 month follow up period
  Length of hospitalization measured in days from the Index Procedure, including days in intensive care unit (ICU) vs. standard in-patient hospitalization
Mean total cost of care per subject | During a 6 month follow up period
  Mean total cost of care per subject including: procedure costs, debridement devices used during the procedure, and inpatient hospital stay from the date of procedure to the date of discharge based on reimbursement fee structure expressed in US dollars, Euros or UK Pounds respectively.
  a. Procedure costs will be based on the cost of an endoscopic retrograde cholangiopancreatography (ERCP) which covers room, X-ray, sedation, personnel, and other materials.
Percent reduction in WON collection volume (cm3) | During a 6 month follow up period
  Assessed by contrast enhanced computed tomography (CECT) scan or magnetic resonance imaging (MRI) (Baseline vs. completion of necrosectomy). Percent reduction in WON collection volume (cm3) as assessed by contrast enhanced computed tomography (CECT) scan or magnetic resonance imaging (MRI) (Baseline vs. completion of necrosectomy).
  1. Endoscopic ultrasound (EUS) may be used for imaging only when a subject is contraindicated for MRI and CECT.
  2. WON collection volume will be measured as follows:
  i. Length = longest diameter in cm/mm in the axial plane (left - right) ii. Width = the longest diameter in cm/mm (frontal - dorsal) in the same axial plane as the length, perpendicular on the longitudinal axis.
  iii. Height = longest diameter in cm/mm on coronal plane (cranial - caudal)
Procedure time | During a 6 month follow up period
  Measured in minutes from the point of per-oral scope insertion to scope removal (scope-in / scope-out).
Debridement time | During a 6 month follow up period
  Measured in minutes from the start of the debridement procedure to completion of the debridement procedure, including time to swap devices.
Subject Quality of Life | During a 6 month follow up period
  Subject quality of life (QOL) as assessed by a SF-36 questionnaire performed at Baseline, Discharge, and at the 1, 3, and 6 Month Post Necrosectomy Follow-up Visits.
The number of device deficiencies, defined as any inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance including malfunction, use errors, and inadequate labelingprocedure | During a 6 month follow up period
  Assessed by the Investigator during each DEN procedure. This may include malfunctions, use error, or inadequacy in the information supplied by the manufacturer

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bruno, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (12):
- United States (3):
  - University of Alabama Medical Center, Birmingham, Alabama
  - California Pacific Medical Center, San Francisco, California
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Copenhagen University Hospital, Hvidovre, Denmark
- Germany (2):
  - Evangelical Hospital, Düsseldorf
  - University of Frankfurt, Frankfurt
- Italy (2):
  - Humanitas Reserach Hospital & Humanitas University, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Netherlands (3):
  - Charlotte van Veldhuisen, Amsterdam
  - Amsterdam University Medical Center, Amsterdam
  - St. Antonius Hospital, Nieuwegein
- Central Manchester University Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No